CLINICAL TRIAL: NCT05526378
Title: Effect of Three Different Sensory Interventions on Pain Level During Heel Blood Collection in Term Infant: a Randomized Controlled Study
Brief Title: Effect of Three Different Sensory Interventions on Pain Level During Heel Blood Collection in Term Infant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elif Dogan, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2022/94
Record Dates: First submitted 2022-08-20; First posted 2022-09-02 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2023-07

CONDITIONS: Infant; Pain
Keywords: infant; pain; mother's milk; mother's voice; skin contact
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group 1 (mother's voice) (Experimental): The mother called her baby between 40 and 60 decibels loudness. The intervention was continued 5 minutes before the heel blood collection and continued until the 5th minute after the procedure. NIPS score was saved in 5 minutes before the heel blood collection and continued until the 5th minute after the procedure.
  Benetech brand GM1352 model decibel meter was used to measure the loudness.
  Interventions: Behavioral: Sensory Interventions
- Group 2 (mother's milk) (Experimental): Breast milk was dripped onto the gauze in an amount to wet the entire 2,5cm*2,5cm sterile gauze. The gauze was then placed close to the baby's nose wings. The intervention was continued 5 minutes before the heel blood collection and continued until the 5th minute after the procedure. NIPS score was saved in 5 minutes before the heel blood collection and continued until the 5th minute after the procedure
  Interventions: Behavioral: Sensory Interventions
- Group 3 (skin to skin contact) (Experimental): Skin-to-skin contact between mother and baby is provided. The intervention was continued 5 minutes before the heel blood collection and continued until the 5th minute after the procedure. NIPS score was saved in 5 minutes before the heel blood collection and continued until the 5th minute after the procedure
  Interventions: Behavioral: Sensory Interventions
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Sensory Interventions — Group 1 will be hear mother's voice before, during and after the procedure. Group 2 will be sniffed mother's breast milk before, during and after the procedure.
  Group 3 will be skin contact with mother's before, during and after the procedure.
  Arms: Group 1 (mother's voice); Group 2 (mother's milk); Group 3 (skin to skin contact)

SUMMARY:
Background: Healthy newborns undergo many painful procedures in the first hours of life. Damage caused by painful procedures can lead to structural and functional changes that can affect adult life. Various non-pharmacological methods have been reported in the literature for pain management. The aim of the study is to investigate the effect of the method that appeals to 3 different senses (mother's voice, breast milk smell, mother's contact) on the level of pain during heel blood collection.

Method: The population of the study consisted of babies who were hospitalized in a hospital's neonatal unit between December 2022 and May 2023 and who heel blood taken. The Neonatal-Infant Pain (NIPS) Scale and data collection form were used to obtain the data. 120 newborns who met the study criteria were randomly divided into group 1 (n=30) , group 2 (n=30), group 3 (n=30), control group (n=30). All intervention was continued 5 minutes before the heel blood collection and continued until the 5th minute after the procedure. The mother called her baby between 40 and 60 decibels loudness for group 1. Breast milk was dripped onto the gauze in an amount to wet the entire 2,5cm*2,5cm sterile gauze and the gauze was then placed close to the baby's nose wings for group 2. Skin-to-skin contact between mother and baby is provided for group 3. NIPS score was saved in 5 minutes before the heel blood collection and continued until the 5th minute after the procedure for all groups.

ELIGIBILITY:
Inclusion Criteria:

* Born between 37+0/7 - 41+6/7 gestational weeks,
* Gestational age and birth weight are compatible,
* Healthy newborns with stable vital signs.

Exclusion Criteria:

* Hearing problems,
* Suction problem
* Congenital anomaly,
* Need hospitalization in the neonatal intensive care unit.

Ages: 24 Hours to 48 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
NIPS scale | Expecting during procedure
  Neonatal Infant Pain Scale (NIPS) consists of 6 items (facial expression, crying, breathing pattern, arms, legs, alertness) and is evaluated between 0-7 points in total. As the score increases, the level of pain increases.
NIPS scale | 5 minutes after procedure
  Neonatal Infant Pain Scale (NIPS) consists of 6 items (facial expression, crying, breathing pattern, arms, legs, alertness) and is evaluated between 0-7 points in total. As the score increases, the level of pain increases.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Dogan, Principal Investigator — Researcher Assistant
Locations (1):
- Istanbul University Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lin CH, Liaw JJ, Chen YT, Yin T, Yang L, Lan HY. Efficacy of Breast Milk Olfactory and Gustatory Interventions on Neonates' Biobehavioral Responses to Pain during Heel Prick Procedures. Int J Environ Res Public Health. 2022 Jan 22;19(3):1240. doi: 10.3390/ijerph19031240. PMID 35162263
- [Background] McPherson C, Miller SP, El-Dib M, Massaro AN, Inder TE. The influence of pain, agitation, and their management on the immature brain. Pediatr Res. 2020 Aug;88(2):168-175. doi: 10.1038/s41390-019-0744-6. Epub 2020 Jan 2. PMID 31896130
- [Background] McNair C, Campbell-Yeo M, Johnston C, Taddio A. Nonpharmacologic Management of Pain During Common Needle Puncture Procedures in Infants: Current Research Evidence and Practical Considerations: An Update. Clin Perinatol. 2019 Dec;46(4):709-730. doi: 10.1016/j.clp.2019.08.006. Epub 2019 Aug 26. PMID 31653304
- [Background] Zhang S, Su F, Li J, Chen W. The Analgesic Effects of Maternal Milk Odor on Newborns: A Meta-Analysis. Breastfeed Med. 2018 Jun;13(5):327-334. doi: 10.1089/bfm.2017.0226. Epub 2018 May 7. PMID 29733222
- [Background] Benoit B, Newman A, Martin-Misener R, Latimer M, Campbell-Yeo M. The influence of breastfeeding on cortical and bio-behavioural indicators of procedural pain in newborns: Findings of a randomized controlled trial. Early Hum Dev. 2021 Mar;154:105308. doi: 10.1016/j.earlhumdev.2021.105308. Epub 2021 Jan 12. PMID 33513546
- [Background] Kucuk Alemdar D, Kardas Ozdemir F. Effects of Having Preterm Infants Smell Amniotic Fluid, Mother's Milk, and Mother's Odor During Heel Stick Procedure on Pain, Physiological Parameters, and Crying Duration. Breastfeed Med. 2017 Jun;12:297-304. doi: 10.1089/bfm.2017.0006. Epub 2017 Apr 17. PMID 28414516
- [Background] Yilmaz D, Yilmaz Kurt F. The effect of foot reflexology on procedural pain before heel lancing in neonates. Arch Pediatr. 2021 May;28(4):278-284. doi: 10.1016/j.arcped.2021.02.015. Epub 2021 Mar 11. PMID 33715931
- [Background] Filippa M, Devouche E, Arioni C, Imberty M, Gratier M. Live maternal speech and singing have beneficial effects on hospitalized preterm infants. Acta Paediatr. 2013 Oct;102(10):1017-20. doi: 10.1111/apa.12356. Epub 2013 Aug 8. PMID 23848529
- [Background] Cakirli M, Acikgoz A. A Randomized Controlled Trial: The Effect of Own Mother's Breast Milk Odor and Another Mother's Breast Milk Odor on Pain Level of Newborn Infants. Breastfeed Med. 2021 Jan;16(1):75-81. doi: 10.1089/bfm.2020.0222. Epub 2020 Oct 20. PMID 33085532
- [Background] Filippa M, Monaci MG, Spagnuolo C, Serravalle P, Daniele R, Grandjean D. Maternal speech decreases pain scores and increases oxytocin levels in preterm infants during painful procedures. Sci Rep. 2021 Aug 27;11(1):17301. doi: 10.1038/s41598-021-96840-4. PMID 34453088
- [Derived] Duman R, Dogan E, Kaya HD, Tepe M. The Effect of Three Different Sensory Interventions (Mother's Voice, Mother's Milk, and Mother's Holding) During Heel Lance on Pain Level in Term Newborns: A Randomized Controlled Trial. Breastfeed Med. 2025 May;20(5):345-352. doi: 10.1089/bfm.2024.0197. Epub 2025 Feb 7. PMID 39918942